CLINICAL TRIAL: NCT03322891
Title: Improving Health Literacy in African-American Prostate Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Viraj Master, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00091879
Record Dates: First submitted 2017-10-23; First posted 2017-10-26 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: Urology
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educational Supplement (Experimental): Participants diagnosed with prostate cancer will receive education for treatment options and treatment side effects.
  Interventions: Other: Educational Supplement; Other: Standard Practice Education

INTERVENTIONS:
Other: Educational Supplement — Participants will receive education about prostate cancer and treatments using models and props during a face-to-face interview. During the interview, participants will also be asked about medical terms and treatments regarding prostate cancer. The interview will last 45 to 60 minutes.
Other: Standard Practice Education — Participants will receive traditional standard of care education regarding prostate cancer treatments and side effects provided by their physician.

SUMMARY:
Investigators propose an observational interview study to explore how patients understand treatment conversations with their physicians within the framework of health literacy. The study team will test whether patients' understanding of treatment options and side effects can be improved when patients receive a low literacy educational supplement after meeting with their urologist. Investigators will interview a group of newly diagnosed, early stage, African American prostate cancer patients.

DETAILED DESCRIPTION:
Investigators propose an observational interview study to explore how patients understand treatment conversations with their physicians within the framework of health literacy. The study team will test whether patients' understanding of treatment options and side effects can be improved when patients receive a low literacy educational supplement after meeting with their urologist. Investigators will interview a group of newly diagnosed, early stage, African American prostate cancer patients.

Investigators hypothesize that the delivery of a scripted, tailored, low literacy educational supplement will result in a statistically significant decrease in decisional conflict, and a statistically significant improvement in comprehension of cancer treatment and its side effects compared to standard practice.

The study team will measure patients' comprehension of treatment options and side effects, as well as decisional conflict; after standard practice, and again after exposure to the educational supplement. Investigators will compare the urologists' assessment of patients' 1) health literacy 2) preferences for side effects 3) stage of decision making, 4) treatment choice or predisposition toward treatment choice. 5) preference for role in decision making (active, passive, or shared with physician); to measures obtained from patients. These comparisons will allow investigators to quantify the potential benefit to the physician of information obtained through the interview and low literacy educational supplement.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone pathology review of their prostate biopsy at Emory University, Grady Memorial Hospital, Saint Joseph's Hospital, and Atlanta VA Medical Center with AJCC clinical stage T1-T2 prostate cancer by physical exam

Exclusion Criteria:

* RN or MD degree
* History of head injury or dementia
* History of cognitive impairment
* Unable to undergo the informed consent process and the study interview in English per the judgment of the primary urologist or urological provider

Ages: 25 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2016-07-21 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Decisional Conflict Scale Score | Baseline, Post-Intervention (Up to 6 Weeks)
  The decisional conflict scale measures personal perceptions of : a) uncertainty in choosing options; b) modifiable factors contributing to uncertainty such as feeling uninformed, unclear about personal values and unsupported in decision making; and c) effective decision making such as feeling the choice is informed, values-based, likely to be implemented and expressing satisfaction with the choice. Scores range from 0 (no decisional conflict) to 100 (extremely high decisional conflict).
Change in Comprehension of Treatment Options Score assessed by Interview | Baseline, Post-Intervention (Up to 6 Weeks)
  Comprehension of treatment options will be scored as dichotomous variables, correct or incorrect. The changes in the proportion of patients who correctly understand treatment after standard practice compared to the proportion who correctly understand treatment after the low literacy supplement will be analyzed.
Change in Comprehension of Side Effects Score assessed by Interview | Baseline, Post-Intervention (Up to 6 Weeks)
  Comprehension of side effects will be scored as dichotomous variables, correct or incorrect. The changes in the proportion of patients who correctly understand side effects after standard practice compared to the proportion who correctly understand treatment after the low literacy supplement will be analyzed.

SECONDARY OUTCOMES:
Rapid Estimate of Adult Literacy in Medicine (REALM) Score | Baseline
  The REALM is a screening instrument to assess an adult patient's ability to read common medical words and lay terms for body parts and illnesses. Scores are assessed on an education grade equivalent;
  0-18 = 3rd Grade and Below Will not be able to read most low literacy materials; will need repeated oral instructions, materials composed primarily of illustrations, or audio or video tapes
  19-44 = 4th to 6th Grade Will need low literacy materials; may not be able to read prescription labels
  45-60 = 7th to 8th Grade Will struggle with most patient education materials
  61-66 = High School Will be able to read most patient education materials
Change in the Stage of Decision Making Scale Score | Baseline, Post-Intervention (Up to 6 Weeks)
  Stage of decision making refers to individual's readiness to engage in decision making, progress in making a choice, and receptivity to considering or re-considering options. This tool is not scored. However, the categories can be used to determine co-variation in decisional conflict (tends to be higher in earlier stages) and success of interventions (success higher among those in active deliberation stage).

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Kilbridge, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Atlanta VA Medical Center, Atlanta, Georgia
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Undecided